CLINICAL TRIAL: NCT00746265
Title: Acceptance-based Behavior Treatment: An Innovative Weight Control
Brief Title: Behavioral Treatment for Weight Loss
Acronym: MYH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21DK080430 (NIH); 1R21DK080430 (NIH)
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Overweight and Obesity
Keywords: behavioral interventions for weight loss
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBT (Active Comparator): Standard behavioral treatment based on the LEARN manual.
  Interventions: Behavioral: Behavioral weight loss intervention
- ABT (Active Comparator): Acceptance-based group that is based on the behavioral interventions contained in LEARN manual
  Interventions: Behavioral: Behavioral weight loss intervention

INTERVENTIONS:
Behavioral: Behavioral weight loss intervention — Participants in both conditions are provided nutritional education and behavioral strategies for weight loss (consistent with the LEARN program). Participants in SBT are taught the cognitive and motivational strategies used in LEARN while participants in ABT are taught acceptance-based strategies (e.g., acceptance, mindfulness).

SUMMARY:
This project compares gold standard cognitive-behavioral therapy (based on LEARN, Diabetes Prevention Program, LOOK Ahead) used in both research and clinical settings, with acceptance-based behavioral therapy for weight loss. Standard behavior treatment (SBT) focuses on modifying eating, thinking, and activity levels. Participants limit their daily caloric intake, keep food records, increase physical activity, and practice weight control behaviors, such as stimulus control, cognitive restructuring, alternative coping skills, and distinguishing hunger from cravings. The acceptance-based approach (ABT) incorporates the behavioral and nutritional components, but replaced the cognitive and motivational components with components that are consistent with an acceptance-based approach, such as acceptance and willingness to experience cravings, cognitive defusion, mindfulness training to interrupt automatic eating, and values work. These components are drawn from Acceptance and Commitment Therapy (ACT; Hayes, Strosahl, & Wilson, 1999), a cognitive-behavioral therapy that has been gaining increasing attention and empirical support (Bach & Hayes, 2002; Bond & Bunce, 2000; Hayes et al. 2004). Though relatively new, acceptance-based strategies have demonstrated effectiveness in helping individuals to respond to unwanted thoughts and feelings (Hayes, Rissett, Korn, Zettle, Rosenfarb, Cooper, & Grundt, 1999, Keogh, Bond, Hanmer, & Tilston, 2005) and offer a novel alternative to control-based strategies (such as distraction and confrontation).

Participants in this study will be randomly assigned to either the traditional behavioral therapy condition (SBT) or the acceptance-based behavioral therapy condition (ABT). Both conditions are delivered in group format. A total of 30, 75 minute sessions will take place over the course of 40 weeks.

Specific Aims

1. To evaluate the feasibility and acceptability of the treatment, and its short and moderate-term effectiveness relative to the current gold standard behavioral treatment (SBT).
2. To evaluate the effectiveness of ABT with novice clinicians and with weight control experts.
3. To evaluate the effectiveness of ABT would be moderated by mood disturbance, emotional eating, disinhibition or susceptibility to food stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 65
* Fluent in English
* Body mass index (BMI) of 25 kg/m2 higher
* Agrees to not join another weight loss program for 9 months

Exclusion Criteria:

* Lactating, pregnant, or planning to become pregnant in the next two years
* Currently taking a medication or having medical/psychiatric problem known to cause weight loss or weight gain (unless medication is long-term and dosage is unchanging - e.g., Synthroid)
* A medical or psychiatric condition that limits ability to comply with the program's behavioral recommendations (including physical activity)
* Current or history in the past ten years of an eating disorder
* Plans to leave the Philadelphia areas within the next nine months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
BMI change | end of treatment and 6 month follow-up

SECONDARY OUTCOMES:
Change in acceptance-based variables (e.g., mindfulness) | end of treatment and 6 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Department of Psychology, 245 N. 15th Street, MS 626, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chabria R, Hagerman CJ, Crane N, Ehmann M, Knudsen FM, Brown KL, Forman E, Butryn ML. Racial disparities in the efficacy of traditional versus acceptance-based behavioral weight loss. Health Psychol. 2025 Jul 24:10.1037/hea0001537. doi: 10.1037/hea0001537. Online ahead of print. PMID 40705619
- [Derived] Forman EM, Manasse SM, Butryn ML, Crosby RD, Dallal DH, Crochiere RJ. Long-Term Follow-up of the Mind Your Health Project: Acceptance-Based versus Standard Behavioral Treatment for Obesity. Obesity (Silver Spring). 2019 Apr;27(4):565-571. doi: 10.1002/oby.22412. Epub 2019 Feb 26. PMID 30806492
- [Derived] Forman EM, Butryn ML, Juarascio AS, Bradley LE, Lowe MR, Herbert JD, Shaw JA. The mind your health project: a randomized controlled trial of an innovative behavioral treatment for obesity. Obesity (Silver Spring). 2013 Jun;21(6):1119-26. doi: 10.1002/oby.20169. Epub 2013 May 13. PMID 23666772